CLINICAL TRIAL: NCT03802357
Title: Effects of Moderate vs. High Intensity Exercise Training During Pulmonary Rehabilitation in Alpha-1 Antitrypsin Deficiency Patients
Brief Title: Effects of Different Exercise Training Modalities in Alpha-1 Antitrypsin Deficiency Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Head physician, Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAT Training
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Chronic Obstructive Pulmonary Disease; Alpha 1-Antitrypsin Deficiency
Keywords: Pulmonary rehabilitation; Exercise training; Alpha-1 Antitrypsin deficiency
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; alpha 1-Antitrypsin Deficiency | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two Intervention Groups (high vs. moderate Training intensity).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High training intensity (Experimental): Exercise Training with high intensities consists of a cycling Interval Training at 100% of the individual Peak work rate, resistance Training for 3 sets à 8 repetitions and squats on a Vibration plate.
  Interventions: Procedure: Exercise training
- moderate training intensity (Active Comparator): Exercise Training with moderate intensities consists of a cycling endurance Training at 60% of the individual Peak work rate, resistance Training for 3 sets à 20 repetitions and squats on the floor.
  Interventions: Procedure: Exercise training

INTERVENTIONS:
Procedure: Exercise training — Patients perform an exercise Training program of 3 weeks Duration including endurance Training, resistance Training and squat Training. This program is part of an inpatient pulmonary Rehabilitation.

SUMMARY:
Pulmonary rehabilitation (PR) including exercise training is highly effective by improving health-related quality of life, exercise capacity and symptoms in patients with chronic obstructive pulmonary disease (COPD). Therefore, PR is a main component in the management of COPD. In a former study patients with Alpha-1 Antitrypsin deficiency (A1ATD)-related COPD (genotype PiZZ) have been found to show smaller improvements in exercise capacity after a 3-week inpatient PR program compared to COPD patients without A1ATD (genotype PiMM)[1]. These between-group differences were mirrored by missing adaptations of the fatigue-resistant skeletal muscle fibre type I in A1ATD patients. This was in contrast to COPD patients without A1ATD who increased the proportion of this fibre type after PR. Myofibre type I is crucial because it enables patients for physical endurance activities (walking, cycling etc.) during their daily life.

The aim of this study is to compare the effects of an exercise Training program with high vs. moderate Training intensity in order to find a Training modality which improves Training effects in A1ATD patients.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients with A1ATD (genotype PiZZ)
* COPD patients without A1ATD (genotype PiMM)
* Global initiative for chronic obstructive lung disease (GOLD) stage III-IV
* Medical Treatment according to recent A1ATD guidelines

Exclusion Criteria:

* General exclusion criteria for physical Training such as acute coronary Syndrome, acute myo- or pericarditis, acute lung embolism, acute heart failure, orthopedic comorbidities which prevent patients from participating in exercise Training program.
* No written informed consent
* Non-compliance

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Endurance shuttle walk test (ESWT) | Change in the duration of the ESWT from day 1 to day 21
  The ESWT is performed at 85% of the Peak gate Speed, measured during the Initial incremental shuttle walk test.

SECONDARY OUTCOMES:
Oxygen saturation | Change in the oxygen saturation at isotime from day 1 to day 21
  Outcome will be assessed at the the time Point of the end of the shortest ESWT ("isotime").
Heart rate | Change in the heart rate at isotime from day 1 to day 21
  Outcome will be assessed at the the time Point of the end of the shortest ESWT ("isotime").
Partial pressure of carbon dioxide (CO2) | Change in the partial pressure of CO2 at isotime from day 1 to day 21
  Parameter will be measured by Sentec (R) device. Outcome will be assessed at the the time Point of the end of the shortest ESWT ("isotime").
Lactate concentration | Change in lactate concentration at isotime from day 1 to day 21
  Outcome will be assessed at the the time Point of the end of the shortest ESWT ("isotime").
Perceived Dyspnea | Change in perceived dyspnea at isotime from day 1 to day 21
  Dyspnea will be rated on a 0 to 10-point BORG scale where lower values represent less dyspnea and vice versa. The total score will be assessed at the the time Point of the end of the shortest ESWT ("isotime").
Strength capacity in knee extension | Change in strength from day 1 to day 21
  Strength will be measured by a Hand Held Dynamometer (Microfet (R)).
Balance performance | Change in balance performance from day 1 to day 21
  absolute path length will be measured on a force plate (Leonardo (R)) during the Tandem stance

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, Prof. Dr., Principal Investigator — Schoen Klinik Berchtesgadener Land
Locations (1):
- Schoen Klinik Berchtesgadener Land, Schönau am Königssee, Germany

IPD SHARING:
Plan to Share IPD: No